CLINICAL TRIAL: NCT04811781
Title: Epidemiological Features and Clinical Course of SARS-CoV-2 Infection in Cancer Patients Within the Veneto Oncology Network: the ROVID Study
Brief Title: Epidemiological Features and Clinical Course of COVID -19 Infection in Cancer Patients: The Rovid Study
Status: Completed | Type: Observational
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: Rovid
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer Patients with SARS-COV-2 infection.

SUMMARY:
The study aims to retrospectively collect epidemiological and clinical data in patients with solid tumors and SARS Covid2 infections belonging to oncology centers within the Veneto Oncology Network

DETAILED DESCRIPTION:
The aim of this study is to create a Veneto Oncology Network with the aim of collecting clinical and epidemiological data of cancer Patients affected by SAR- Covid-2 infection over a period of 1 year. Descriptive statistical approaches will be used to process the data.

The aim is to evaluate the development rate of severe clinical forms of infection in patients with SARS-Cov-2 and the possible association with tumour characteristics and treatment.

In addition, the results of serological tests can be compared with the outcome of the diagnostic swabs and the clinical evolution of the infection in order to obtain more information regarding the significance of specific antibody development.

ELIGIBILITY:
Inclusion Criteria:

* be 18 Years and older
* cancer patients belonging to Veneto 's Oncological Network
* Patients with SAR COV-2 infection

Exclusion Criteria:

* Patients with no SAR COV2 Infection
* Volunteers
* No Cancer Patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with SAR COV-2 infection within the Veneto Oncology Network
Sampling Method: Non-Probability Sample
Enrollment: 761 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
The rate of SAR-COV2 infection development in association with tumor characteristics. | through study completion, an average of 18 months.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - istituto Oncologico Veneto -UOSD Melanoma, Padua, PD
  - Aulss1 Dolomiti, Belluno
  - Istituto Oncologico Veneto -UOC Oncologia 1, Padua